CLINICAL TRIAL: NCT03652155
Title: Evaluating the Relationship Between Hard and Soft Tissue Advancement in Orthognathic Surgery
Status: Completed | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: 7694
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Dentofacial Deformities
MeSH Terms: conditions — Dentofacial Deformities | interventions — Orthognathic Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthognathic Surgery Patients: The study cohort will be patients undergoing orthognathic surgery for correction of an existing dentofacial deformity.
  Interventions: Procedure: Orthognathic surgery

INTERVENTIONS:
Procedure: Orthognathic surgery — Patient's pre and post operative hard and soft tissues will be evaluated retrospectively through the use of con-beam computed tomography imaging for hard tissue evaluation and 3DMd three dimensional photography for soft tissue imaging.

SUMMARY:
This study aims to evaluate the relationship between hard and soft tissue advancement during orthognathic surgery. The use of typical pre and post operative imaging consisting of con-beam computed tomography will be used, in conjunction with a 3D camera to evaluate hard and soft tissue points before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient's undergoing orthognathic surgery for correction of a dentofacial deformity

Exclusion Criteria:

* patients with previous orthognathic surgery patients with cranio-facial syndromes

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Any patient undergoing orthognathic surgery for correction of a pre-existing dentofacial deformity.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Hard and soft tissue change | pre operative and post operative imaging is taken immediately before, and 24 hours post operatively, respectively.
  The difference between standard pre and post operative hard and soft tissue positioning will be evaluated. Comparisons will be made between the actual bony advancement of a particular bony landmark, and compare that advancement to the advancement seen with a corresponding soft tissue landmark.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
This data will not be available to other researchers.